CLINICAL TRIAL: NCT04397887
Title: Seminal TEX101 as a Predictor of Recovery of Spermatogenesis in Azoospermic Men With Palpable Varicocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Wael Ragab, Andrology consultant/ lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CairoU Azoospermia Vx TEX101
Record Dates: First submitted 2020-05-07; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Azoospermia, Nonobstructive; Varicocele
Keywords: Varicocele; Azoospermia; TEX 101
MeSH Terms: conditions — Azoospermia, Nonobstructive; Varicocele; Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men with Azoospermia and varicocele (Experimental): In this single arm study, TEX 101 is measured in the seminal fluid of all participants, and it will be used as a predictor for appearance of sperms in the ejaculate in 3 and 6 moths follow-up periods
  Interventions: Procedure: micro-surgical varicocelectomy

INTERVENTIONS:
Procedure: micro-surgical varicocelectomy — Sub-inguinal micro-surgical varicocelectomy

SUMMARY:
The aim of the study is to assess if seminal TEX 101 can predict the restoration of spermatogenesis and appearance of sperms in the ejaculate after micro-surgical varicocelectomy among azoospermic patients.

DETAILED DESCRIPTION:
Male patients (40) cases attending the outpatient clinic of Andrology at KASR EL-AINI university hospitals, all patients presented with azoospermia, age:18-43 years, complaining mainly of infertility or accidently discovered azoospermia during premarital check-up or chronic testicular pain caused by longstanding varicocele. Infertile Non Obstructive Azoospermia (NOA) (n=40) subjected to varicocelectomy and patients evaluated 3 months after varicocelectomy by semen analysis, then according to results population divided into 2 groups: Group A (Responders): Patients with positive semen analysis for

sperms 3 months after varicocelectomy.

Group B (Non Responders): Patients with no sperms in semen analysis

in 3 and/or 6 months after varicocelectomy.

Method of Estimation of human TEX101 in semen:

A 1 ml collected semen samples were centrifuged for 20 minutes at 1000xg at 4 o C, then supernatant of each sample was collected for estimation of TEX101. The human TEX101 (Testis expressed 101) was assayed by commercially available ELISA kit supplied by Wuhan Fine Biotech Co., Ltd. China.

Principle of the procedure:

This kit was based on sandwich enzyme-linked immune-sorbent assay technique. Anti- TEX101 antibody was pre-coated onto 96-well plate. The biotin conjugated antibody was used as detection antibodies. The standards, test samples and biotin conjugated detection antibody were added to the wells subsequently, and washed with wash buffer.

HRP-Streptavidin was added and unbound conjugates were washed away with wash buffer. TMB substrates were used to visualize HRP enzymatic reaction. TMB was catalyzed by HRP to produce a blue color product that changed into yellow after adding acidic stop solution. The intensity of yellow is proportional to the target amount of sample captured in plate.

ELIGIBILITY:
Inclusion Criteria:

* Azoospermia in at least 2 separate semen analyses
* Palpable varicocele

Exclusion Criteria:

* Obstructive azoospermia
* Abnormal Karyotype
* Previous chemotherapy, radiotherapy and or diagnosed maligancy.
* previous testicular of inguinal surgeries.
* secondary azoospermia

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Sperm retrieval in ejaculate | 3 months follow-up
  finding sperms in the ejaculate
Sperm retrieval in ejaculate | 6 months follow-up
  finding sperms in the ejaculate

CONTACTS AND LOCATIONS:
Locations (1):
- Andrology department, Faculty of Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No